CLINICAL TRIAL: NCT06460714
Title: Effects of Shockwave Therapy on Crouched Gait and Hamstring Flexibility in Children With Diplegic Cerebral Palsy.
Brief Title: Effects of Shockwave Therapy on Crouched Gait Due to Hamstring Flexibility in Cerebral Palsy Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0775
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Shock wave; Hamstring flexibility; Crouched gait
MeSH Terms: conditions — Cerebral Palsy | interventions — Extracorporeal Shockwave Therapy; Orthotic Devices

STUDY DESIGN:
Intervention Model Description: Randomized Control trial in which non-probability convenient sampling will be used. Both group of spastic CP of age 6 to 12 will be randomly divided. Group A will receive shockwave, stretching and orthosis. Group B will receive stretching and orthosis.
Who Masked: Participant
Masking Description: Participants will get separated treatment protocols and possible efforts will be put to mask the both groups about the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shock wave therapy, stretching and orthosis (Experimental): Shortwave therapy, stretching and orthotics will be provided to Group A. Shock wave session will be provided for 20 minutes thrice a week. Five days in a week provided five minutes with 30 seconds sustained stretch will be provided and than orthotics will be used to obtained the sustained effect.
  Interventions: Other: Shock wave therapy, stretching and orthosis
- Stretching, strengthening and orthosis (Active Comparator): In Group B spastic diplegic children just given stretching with strengthening and orthotics. We provide sustained 30 seconds stretch with 30 seconds rest for 5 minutes and followed with forty repetition of hip flexor and knee flexors and range will be maintained by applying orthosis.
  Interventions: Other: Stretching, strengthening and orthosis

INTERVENTIONS:
Other: Shock wave therapy, stretching and orthosis — Shortwave therapy, stretching and orthotics will be provided to Group A. Shock wave session will be provided for 20 minutes thrice a week. Five days in a week provided five minutes with 30 seconds sustained stretch will be provided and than orthotics will be used to obtained the sustained effect.
  Arms: Shock wave therapy, stretching and orthosis
Other: Stretching, strengthening and orthosis — In Group B spastic diplegic children just given stretching with strengthening and orthotics. We provide sustained 30 seconds stretch with 30 seconds rest for 5 minutes and followed with forty repetition of hip flexor and knee flexors and range will be maintained by applying orthosis.
  Arms: Stretching, strengthening and orthosis

SUMMARY:
Randomized controlled trial will be conducted on thirty-two cerebral palsy children in Punjab Special School. Spastic Diplegic CP children with GMFCs level III, IV, V with age range of 6 to 12. These children have limited range of hamstring muscles. Assessment will be measured Pre and Post treatment by goniometer of crouched gait in standing and lying on couch. Crouched gait will be measured by Knee flexion in standing and lying. To measure hamstring flexibility ROM of knee extension is measured with 90 flexion at hip joint. Spasticity in this study will be assessed by GMFM-88 and modified Ashworth scale.

DETAILED DESCRIPTION:
Shortwave therapy, stretching and orthotics will be provided to Group A. Shock wave session will be provided for 20 minutes thrice a week. Five days, five minutes with 30 seconds sustained stretch will be provided and than orthotics will be used to obtained the sustained effect.

In Group B spastic diplegic children just given stretching with strengthening and orthotics. We provide sustained 30 seconds stretch with 30 seconds rest for 5 minutes and followed with forty repetition of hip flexor and knee flexors and range will be maintained by applying orthosis.

ELIGIBILITY:
Inclusion Criteria:

* Children with GMFCS level I, II & III.
* Passive range of motion of knee extension is limited to 20 degree with hip 90 degree.
* Age between 6 to 12 years.

Exclusion Criteria:

* Children with epileptic history
* Previous muscular lengthening technique applied
* Previous history of botox injection used.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2024-04-05 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
Modified Ashwarth Scale | 8 weeks
  The Modified Ashworth Scale (MAS) is a commonly used clinical assessment tool to evaluate muscle tone and spasticity in individuals with neurological conditions such as spastic cerebral palsy. It is a reliable and valid method for grading muscle resistance during passive movement. interrater reliability of AS and MAS varied from moderate to good. ICC scores of AS were between 0.54 and 0.78 and MAS were between 0.61-0.87. Test-retest results of AS and MAS varied from poor to good. ICC values were between 0.31 and 0.82 for AS and between 0.36 and 0.83 for MAS
GMFM-88 | 8 weeks
  The Gross Motor Function Measure-88 (GMFM-88) is widely used tool for assessing changes in gross motor function among children with cerebral palsy. It comprising 88 items across five domains. GMFM-A includes activities such as lying and rolling, GMFM-B includes sitting, Crawling and kneeling includes in GMFM-C, GMFM-D includes standing and walking, running and jumping includes in GMFM-E. The reliability of GMFM-88 is 0.75 to 1.0.
Goniometer | 8 weeks
  A goniometer is a measurement tool commonly used in rehabilitation and physical therapy to assess the range of motion (ROM) of various joints in the body. It consists of a stationary arm and a movable arm with a protractor-like scale, allowing for precise measurement of joint angles. By aligning the stationary arm with the joint's axis and the movable arm with the body segment, the goniometer provides objective measurements of joint flexibility, mobility, and muscle strength. The goniometer provides valuable quantitative data that can guide treatment planning, monitor patient progress, and assess functional outcomes related to joint movement and mobility.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Fahad Asif, MS*, Principal Investigator — Riphah International University
Locations (1):
- Punjab Special School, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vitrikas K, Dalton H, Breish D. Cerebral Palsy: An Overview. Am Fam Physician. 2020 Feb 15;101(4):213-220. PMID 32053326
- [Background] Lowing K, Arredondo YC, Tedroff M, Tedroff K. Introduction of the gross motor function classification system in Venezuela--a model for knowledge dissemination. BMC Pediatr. 2015 Sep 4;15:111. doi: 10.1186/s12887-015-0433-5. PMID 26341265
- [Background] Armand S, Decoulon G, Bonnefoy-Mazure A. Gait analysis in children with cerebral palsy. EFORT Open Rev. 2016 Dec 22;1(12):448-460. doi: 10.1302/2058-5241.1.000052. eCollection 2016 Dec. PMID 28698802